CLINICAL TRIAL: NCT05064956
Title: An Open Label, Phase 2 Study to Evaluate the Safety and Immunogenicity of an Ad26.ZEBOV Booster Dose in Human Immunodeficiency Virus Positive (HIV+) Adults Previously Vaccinated With the Ad26.ZEBOV, MVA-BN-Filo Vaccine Regimen
Brief Title: Ad26.ZEBOV Booster in HIV+ Adults Previously Vaccinated With Ad26.ZEBOV/MVA-BN-Filo (EBOVAC HIV+ Booster Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAC52150EBL2010
Record Dates: First submitted 2021-09-15; First posted 2021-10-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2021-08

CONDITIONS: Ebola Virus Disease; Ebola; Hiv
Keywords: Ebola; Vaccine; HIV; Safety; Immunogenicity
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ad26.ZEBOV (Experimental): Ad26.ZEBOV will be given as a booster dose to all participants approximately 4 years after administration of the 2-dose Ebola regimen, Ad26.ZEBOV/MVA-BN-Filo, as part of the parent trial VAC52150EBL2002.
  Interventions: Biological: Ad26.ZEBOV

INTERVENTIONS:
Biological: Ad26.ZEBOV — Ad26.ZEBOV is a non-replicating, monovalent vaccine expressing the full-length Mayinga glycoprotein (GP) of the Ebola virus (formerly known as Zaire ebolavirus), and is produced in human cell line.
  Participants will receive a 0.5mL intramuscular injection of Ad26.ZEBOV, at a concentration of 1x10^11 vp/mL, into the anterolateral deltoid muscle.
  Other Names: Zabdeno®

SUMMARY:
This is an open label study to evaluate the safety and immune response to a booster dose of Ad26.ZEBOV Ebola vaccine in HIV+ adults from Kenya and Uganda. Only participants who have received the 2-dose Ebola vaccine regimen "Ad26.ZEBOV/MVA-BN-Filo " in the VAC52150EBL2002 vaccine trial about 4 years ago are eligible to take part.

Approximately 50 healthy HIV+ adults, aged 18 - 50 years at the time of the parent trial, will be invited. Participants will first be asked to provide consent to participate in this study. Upon receiving the booster vaccination, participants will be followed up for approximately 28 days (+/- 3 days) to collect information on side effects and provide blood samples for antibody measurement.

This study is designed to provide descriptive information regarding vaccine safety and immunogenicity. There is no formal treatment comparisons and no formal testing of statistical hypothesis.

DETAILED DESCRIPTION:
TITLE

An open label, Phase 2 study to evaluate the safety and immunogenicity of an Ad26.ZEBOV booster dose in Human Immunodeficiency Virus positive (HIV+) adults previously vaccinated with the Ad26.ZEBOV, MVA-BN-Filo vaccine regimen.

RATIONALE

In previous Phase 2 and 3 trials, HIV+ adult participants were vaccinated with a 2-dose Ebola vaccine regimen of adenovirus serotype 26 expressing the Ebola virus Mayinga glycoprotein (Ad26.ZEBOV) followed by Modified Vaccinia Ankara Bavarian Nordic vector expressing multiple filovirus proteins (MVA-BN-Filo). This Ebola vaccine regimen elicited humoral immune responses in HIV+ adults comparable to those in HIV-negative adults 21-days after dose 2. However, the durability of vaccine-induced humoral responses was not known.

PRIMARY OBJECTIVES

* To assess the safety and tolerability of a Ad26.ZEBOV booster dose in HIV+ adults previously vaccinated with the Ad26.ZEBOV, MVA-BN-Filo vaccine regimen.
* To assess humoral responses induced by the booster dose against EBOV glycoprotein (GP), as measured by Filovirus Animal Non-Clinical Group (FANG) Enzyme-Linked Immunosorbent Assay (ELISA) at 7 and 21 days.

STUDY DESIGN

This is an open label study to evaluate the immune response to a booster dose of Ad26.ZEBOV administered to HIV+ participants who previously received the 2-dose Ebola vaccine regimen with Ad26.ZEBOV followed by MVA-BN-Filo 28 days or 56 days later in the VAC52150EBL2002 vaccine trial. The Ad26.ZEBOV will be administered as a booster dose in this population approximately 4 years from the time participants received MVA-BN-Filo. Approximately 50 HIV+ adult participants, aged 18 - 50 years at randomisation in the parent trial, VAC52150EBL2002, from Kenya and Uganda will be invited to participate in this trial. Subjects will be asked to consent to participate in this study. Upon receiving the booster vaccination, participants will be followed up for immunogenicity and safety for approximately 28 days (+/- 3 days).

SUBJECT POPULATION

Participants must be healthy (based on physical examination, medical history, and clinical judgment) HIV+ adults who participated in the VAC52150EBL2002 trial. Participants will have to be virologically suppressed and immunologically controlled on highly active antiretroviral therapy (HAART) regimen (HIV viral load < 50 copies/millilitres (mL) and CD4+ T cell count >/= 350 cells/microlitres (uL) within 28 days of study vaccination). The study will be conducted at VAC52150EBL2002 sites in Kenya and Uganda.

PROHIBITIONS AND RESTRICTIONS

1. Travel to an area with active Ebola outbreak during the study period
2. Sexually active female subjects of childbearing potential should use adequate birth control measures from at least 14 days before and 28 days after vaccination
3. No disallowed concomitant therapies are being used

INVESTIGATIONAL PRODUCT, DOSAGE AND ADMINISTRATION

Ad26.ZEBOV is a replication-incompetent monovalent vaccine against Ebola. It consists of an adenovirus serotype 26 vector expressing the full-length Ebola virus (EBOV, formerly known as Zaire ebolavirus) Mayinga GP. A single dose of Ad26.ZEBOV at a dose of 5x10^10 viral particles (vp) will be administered intramuscularly.

SAFETY EVALUATIONS

Solicited local (i.e. injection site) and systemic adverse events (AEs) will be assessed on the day of vaccination and using a diary for a period of seven days following the booster vaccination. Unsolicited adverse events will be tracked for 28 days following booster vaccination, while serious adverse events will be tracked for the duration of the study. The Principal Investigators, together with the sponsor's medical safety officer, will be responsible for the safety monitoring of the study.

Solicited local AEs to be collected in this study include:

* Injection Site Tenderness
* Injection Site Erythema
* Injection Site Swelling
* Itching

Solicited systemic AEs to be collected in this study include:

* body temperature
* fatigue/malaise
* chills
* headache
* nausea/vomiting
* muscle pain
* joint pain

IMMUNOGENICITY EVALUATIONS

Blood will be drawn for assessments of immune responses at Day 1 (prior to vaccination), Day 8 and Day 22. The site staff will perform sample collection and processing according to current versions of approved standard operating procedures.

Future scientific research may be conducted to further investigate Ebola vaccine- and disease-related questions and to study other infections of public health importance in Kenya and Uganda, and neighboring countries. This may include the development of new, or the improvement of existing, techniques to characterise EBOV-directed immune responses or diagnostic tests. No additional samples will be taken for these analyses, however, residual samples from the study tests may be retained for these purposes and analysed after the end of the study.

INDEPENDENT DATA AND MONITORING COMMITTEE (IDMC)

The safety of the Ad26.ZEBOV vaccine has already been shown in HIV+ adults in previous studies. Therefore, the role of the IDMC will be designated to an Independent Medical Reviewer (IMR) to provide medical oversight and detect trends in safety signals. The IMR will periodically review the safety data collected and call for ad hoc safety meetings should any of the pre-specified pausing rules are met or in any situation that could affect participant safety.

PAUSING RULES

1. Death of a participant, considered related to study vaccine or if the causal relationship to the study vaccine cannot be excluded; OR
2. One or more participants experience an serious adverse event (SAE; solicited or unsolicited) that is determined to be related to study vaccine; OR
3. One or more participants experience anaphylaxis or generalised urticaria within 24 hours of vaccination, clearly not attributable to other causes than the study vaccine.

QUALITY ASSURANCE (QA) AND MONITORING

Systematic QA and monitoring of study activities during the clinical study will serve to assure the data reliability and validity, as well as ensure the close adherence to the protocol, Good Clinical Practice (GCP) and contribute to protecting the participant's safety. Automatic data queries will be generated by the Sponsor Data Manager. These queries will be posted in the electronic Data Capture system or sent to the site Investigators via email, if necessary. The QA Committee and external monitors will periodically review these queries and follow up with the sites to ensure resolution. External monitors will also conduct on-site monitoring visits to perform 100% source document verification.

ELIGIBILITY:
Inclusion Criteria:

1. Must have previously received the 2-dose Ebola vaccine regimen in Kenya or Uganda in Cohort 2a of the VAC52150EBL2002 study.
2. Must be aged 18 - 50 years at time of randomisation in the VAC52150EBL2002 study.
3. Must consent to participate in the study by signing or thumbprinting an informed consent form (ICF), indicating that the participant understands the purpose and procedures of the study, as well as the potential risks and benefits of participation.
4. Must be willing/able to ensure that participants adhere to the prohibitions and restrictions specified in this protocol
5. Must be available and willing to participate for the duration of the study visits.
6. Must be in reasonably good medical condition (absence of acquired immunodeficiency syndrome [AIDS]-defining illnesses or clinically significant disease)
7. Must be on a stable regimen of HAART, with a HIV viral load of <50 copies/mL and a CD4+ T-cell count of >350 cells/µL at screening. Must be willing to continue HAART throughout the study.
8. Potential participants must be healthy on the basis of clinical laboratory tests performed at screening.
9. Female subjects of childbearing potential must use adequate birth control measures consistent with local regulations, from at least 14 days before vaccination until the end of the study. Must have a negative pregnancy test at screening and immediately prior to vaccination.
10. Must have a means to be contacted

Exclusion Criteria:

1. Participants in the VAC52150EBL2002 trial who were not in the Cohort 2a, or were allocated to the placebo arm.
2. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products, chicken or egg proteins and aminoglycosides (e.g. gentamicin).
3. Presence of acute illness or axillary temperature ≥38ºC on the day of vaccination. Participants with such symptoms will be deferred.
4. Women who are breast-feeding or known to be pregnant or planning to become pregnant during the study.
5. Clinically significant history of skin disorder, allergy, symptomatic immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, neurological illness.
6. Received a blood transfusion or other blood products within 8 weeks of enrolment.
7. Potential participants who have been vaccinated with live-attenuated vaccines within 30 days before and after the study vaccination, and with inactive vaccine within 15 days before and after the study vaccination.
8. Receipt of any disallowed therapies before the planned administration of the study vaccine.
9. Subjects who, in the opinion of the investigator, are unlikely to adhere to the requirements of the study or are unlikely to complete the study.
10. Any other finding which, in the opinion of the investigator, would increase the risk of an adverse outcome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited adverse events | From the day of the booster to 7 days post-booster vaccination
  Number and percentage of participants with solicited adverse events at the local injection site and systemically
Incidence of unsolicited adverse events | From the day of the booster to 28 days post-booster vaccination
  Number and percentage of participants with any untoward medical event
Vaccine-induced humoral immune responses to the Ebola virus glycoprotein (EBOV GP) | At Day 1 (vaccination)
  EBOV GP antibody concentration measured by FANG ELISA in ELISA Units (EU) per mL.
Vaccine-induced humoral immune responses to the Ebola virus glycoprotein (EBOV GP) | At Day 8
  EBOV GP antibody concentration measured by FANG ELISA in ELISA Units (EU) per mL.
Vaccine-induced humoral immune responses to the Ebola virus glycoprotein (EBOV GP) | At Day 22
  EBOV GP antibody concentration measured by FANG ELISA in ELISA Units (EU) per mL.

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit; Omu Anzala, PhD, Principal Investigator — KAVI - Institute of Clinical Research; Deborah L Watson-Jones, PhD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (2):
- KAVI - Institute of Clinical Research, Nairobi, Kenya
- MRC/UVRI and LSHTM Uganda Research Unit, Masaka, Buganda, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The rights of study subjects and partners, the sharing of data between partners and the transfer of data to external third party will be governed by the Data Sharing Agreement. Deidentified participant-level data collected in this trial will be disseminated through a data repository, such as the Data Compass, that complies with the principles of findability, accessibility, interoperability and reusability (FAIR).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Start date: within 12 months of the study completion date End date: 60 months after the sharing start date Sharing period: 5 years
Access Criteria: Study documents, such as the full protocol, statistical codes, Statistical Analytical Plan, Analytic Code, Independent Medical Reviewer's Terms of Reference, will be available upon request by email to Deborah Watson-Jones (Chief Investigator, Deborah.watson-jones@lshtm.ac.uk), Philip Ayieko (Study Statistician, philip.ayieko@lshtm.ac.uk) or Edward Choi (Study Coordinator, edward.choi@lshtm.ac.uk).
URL: https://datacompass.lshtm.ac.uk/

REFERENCES:
- [Derived] Man-Lik Choi E, Abu-Baker Mustapher G, Omosa-Manyonyi G, Foster J, Anywaine Z, Musila Mutua M, Ayieko P, Vudriko T, Ann Mwangi I, Njie Y, Ayoub K, Mundia Muriuki M, Kasonia K, Edward Connor N, Florence N, Manno D, Katwere M, McLean C, Gaddah A, Luhn K, Lowe B, Greenwood B, Robinson C, Anzala O, Kaleebu P, Watson-Jones D; EBL2010 Study Team. Safety and immunogenicity of an Ad26.ZEBOV booster vaccine in Human Immunodeficiency Virus positive (HIV+) adults previously vaccinated with the Ad26.ZEBOV, MVA-BN-Filo vaccine regimen against Ebola: A single-arm, open-label Phase II clinical trial in Kenya and Uganda. Vaccine. 2023 Dec 7;41(50):7573-7580. doi: 10.1016/j.vaccine.2023.10.055. Epub 2023 Nov 18. PMID 37981473